CLINICAL TRIAL: NCT04069065
Title: Multi Center, Non-comparative, Phase IV Study to Evaluate the Efficacy and Safety of Conversion to TacroBell SR Cap.(Once-Daily Tacrolimus) in Patients Undergoing Maintenance Therapy With Twice-Daily Tacrolimus After Liver Transplantation.
Brief Title: Efficacy and Safety of Once-Daily Tacrolimus in Liver Transplant Recipients (SOUL)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B93_03LT1901
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Liver Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conversion to Once-daily Tacrolimus (Experimental): Conversion to TacroBell slow-release cap.(Once-daily Tacrolimus) at least one year after liver transplantation
  Interventions: Drug: Conversion to Once-daily Tacrolimus

INTERVENTIONS:
Drug: Conversion to Once-daily Tacrolimus — * Orally, once-daily in the morning
  * The first dose is converted to approximately 100% of the existing daily dose, taking into account the subject's blood concentration, after which the investigator check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 3~10ng/ml.
  Other Names: TacroBell slow-release cap.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of conversion to TacroBell slow-release cap.(Once-daily Tacrolimus) in patients undergoing maintenance therapy with Twice-Daily Tacrolimus after liver transplantation.

DETAILED DESCRIPTION:
This study is a multi-center, non-comparative, and phase IV clinical trial that evaluates the efficacy and safety of conversion to TacroBell slow-release cap.(Once-daily Tacrolimus) in patients who have undergone at least one year after liver transplantation and receive maintenance therapy with Twice-Daily Tacrolimus.

Enrolled subjects will take TacroBell slow-release cap.(Once-daily Tacrolimus) for 24 weeks and will conduct scheduled tests with four additional visits.

ELIGIBILITY:
Inclusion Criteria:

* At least one year after liver transplantation
* Over 20 years old(male or female)
* Patient taking tacrolimus twice daily as a maintenance therapy
* Patients with Tacrolimus blood levels of 3-10 at screening
* Agreement with written informed consent

Exclusion Criteria:

* Previously transplanted another organs other than the liver or at the same time
* Diagnosed and clinically treated with acute rejection within the last 6 months
* Patients who have changed the method of administering concomitant immunosuppressants or steroids within the last month
* Diagnosed with cancer in the last five years [Patients, however, who have recovered from skin cancer (squamous cell/basal cell carcinoma) or thyroid cancer, hepatocellular carcinoma without main vessel invasion or extrahepatic metastasis can be enrolled]
* Patients who have positive HIV test result
* Severe systemic infection requiring treatment
* At screening

  * White blood cell count < 1,500/mm^3, or platelet < 50,000/mm^3, or Serum-C r> 2.0mg/dl
  * Liver function test(T-bilirubin, aspartate aminotransferase, alanine aminotransferase)is over 3 times than upper normal limit
* Patients Taking HCV(hepatitis C virus) Therapeutic Drugs
* Pregnant women or nursing mothers
* Fertile women who not practice contraception with appropriate methods
* Participated in other trial within 4 weeks
* In investigator's judgment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-02-22 (Estimated); Study Completion 2021-04-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite efficacy failure | until 24 weeks
  composite efficacy failure include biopsy-confirmed acute rejection, graft loss, death, or follow-up failure

SECONDARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection | until 24 weeks
  episode of biopsy-confirmed acute rejection until 24weeks after conversion
Pathological results of acute rejection | until 24 weeks
  acute rejection using Banff 2016 Criteria and RAI(Rejection activity index) score; total 0~9
Survival rate of transplanted organ | at 24 weeks
Survival rate of Patients | at 24 weeks
Serum-Cr, eGFR(estimated glomerular filtration rate) | at 24 weeks
  eGFR using MDRD(Modification of Diet in Renal Disease) method
Evaluate safety of TacroBell SR. cap. from number of participants with adverse events | until 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea